CLINICAL TRIAL: NCT02646605
Title: Prevalence of Depression Amongst HIV Positive Patients Attending ART Clinic at Lighthouse Clinic, Lilongwe
Brief Title: Depression Amongst HIV Positive Patients in Lilongwe
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Fogarty AIDS international training research program (Unknown)
Responsible Party: Principal Investigator, Mina Hosseinipour, MD, MPH, Clinical Director, University of North Carolina, Chapel Hill
Other Study IDs: 12-2158
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: HIV; AIDS
Keywords: Depression; AIDS; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients initiating ART: HIV positive men and women initiating ART
  Interventions: Other: depression screening
- patients on established ART: HIV positive men and women on established ART
  Interventions: Other: depression screening

INTERVENTIONS:
Other: depression screening — Patient Health Questionnaire

SUMMARY:
Quantitative, validated tools of depression screening will be used to collect data to determine the prevalence of depression and its association with antiretroviral (ARV) adherence amongst HIV positive patients attending ART clinic at Lighthouse Lilongwe, Malawi.

DETAILED DESCRIPTION:
Preliminary data on prevalence and associations will be collected from 200 HIV positive adult men and women attending ART clinic at the Lighthouse in Lilongwe, Malawi. Quantitative, validated tools of depression screening will be used. A short structured demographic questionnaire will be used to collect demographic data. For depression, a Patient Health Questionnaire (PHQ) will be used while alcohol use will be assessed by Alcohol Use Disorders Identification Test (AUDIT) screening tool. The data collected will provide baseline data planning, program development and evaluation, and to promote comprehensive care provision for the people living with AIDS attending ART clinics in Malawi.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* HIV positive men and women accessing care at LH
* Both ART naïve and on ART
* Registered with LH
* Receiving primary care and/ or ART from LH

Exclusion Criteria:

* Too sick to comprehend consent or requiring admission
* Known mentally ill patient on psychiatric drugs
* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women accessing HIV care at Lighthouse clinic, Lilongwe, Malawi will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of depression amongst HIV positive patients attending ART clinic at Lighthouse Lilongwe, Malawi | enrollment
  the survey will be administered one time

CONTACTS AND LOCATIONS:
Overall Officials: Mina Hosseinipour, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lighthouse Clinic, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malawi Demographic Profile 2012
- [Background] Mwale M.C. et al (2006) The Prevalence Of Psychological Distress And Associated Factors Among People Living With Aids Attending Antiretroviral Therapy Clinics In Mzuzu, Malawi: A Cross Sectional Descriptive study. Accessed on 09 June 2012 from www.medcol.mw/mph/.../Charles%20M%20%20Mwale.pdf
- [Background] Guilbert JJ. The world health report 2002 - reducing risks, promoting healthy life. Educ Health (Abingdon). 2003 Jul;16(2):230. doi: 10.1080/1357628031000116808. No abstract available. PMID 14741909
- [Background] Rochon PA, Mashari A, Cohen A, Misra A, Laxer D, Streiner DL, Dergal JM, Clark JP, Gold J, Binns MA. Relation between randomized controlled trials published in leading general medical journals and the global burden of disease. CMAJ. 2004 May 25;170(11):1673-7. doi: 10.1503/cmaj.1031006. PMID 15159365
- [Background] World Health Organisation. (2005). Promoting Mental Health: concepts, emerging evidence, practice: report of the world health organisation, Dept of Mental Health and Substance Abuse in collaboration with the Victorian Health Promotion Foundation & the University of Melbourne. Geneva: World Health Organisation.